CLINICAL TRIAL: NCT03963921
Title: Multicenter, Open-label, Safety and Tolerability Study of Ascending Doses of HepaStem in Patients With Cirrhotic and Pre-cirrhotic Non-alcoholic Steato-hepatitis (NASH)
Brief Title: Safety and Tolerability of HepaStem in Patients With Cirrhotic and Pre-cirrhotic NASH Patients
Acronym: PANASH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP201
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F4 patient population (Experimental): A total of 2 doses are planned to be administered as single or repeated infusions in an ascending manner:
  Interventions: Drug: HepaStem
- F3 patient population (Experimental): A total of 2 doses are planned to be administered as single or repeated infusions in an ascending manner:
  Interventions: Drug: HepaStem

INTERVENTIONS:
Drug: HepaStem — Heterologous human adult liver-derived progenitor cells

SUMMARY:
Multicenter, open-label, safety and tolerability study of ascending doses of HepaStem in patients with cirrhotic and pre-cirrhotic non-alcoholic steato-hepatitis (NASH) to determine the safety and tolerability of ascending single and repeated doses of HepaStem administered to patients with cirrhotic and pre-cirrhotic non-alcoholic steato-hepatitis (NASH)

ELIGIBILITY:
Main Inclusion Criteria:

* Able and willing to provide written informed consent and comply with the requirements of this study protocol
* Age 18 to 70-years old, inclusive
* Proven diagnosis of NASH based on histological evidence from biopsy performed within 6 months for F3 patients and within 2 years for F4 patients prior to Screening If no biopsy is available within these time windows, a biopsy should be performed at Screening NB: For F4 patients for whom the biopsy cannot confirm the diagnosis of NASH, any other causes of underlying liver diseases should be excluded

Main Exclusion Criteria:

* Alcoholic liver disease or alcohol consumption exceeding the daily intake of 140g/w (two doses) for women and of 210g/w (three doses) for men
* Other causes of liver disease including, but not limited to, alcoholic liver disease, active hepatitis B (HbsAg+), hepatitis C (PCR positive), autoimmune disorders, drug-induced hepatotoxicity, Wilson disease, hemochromatosis, and alpha-1-antitryspin deficiency based on medical history and/ or clinical and biological assessment
* Recent recurrent or ongoing thrombotic or bleeding events within 3 months prior the screening
* Patients considered at persistent risk of thrombosis or bleeding at the time of screening
* Patients with high risk of Gastro intestinal bleeding at time of the screening.
* Cerebrovascular, myocardial, or limb arterial thrombotic event within 12 months prior to the screening and/or not considered stabilized by the investigator
* Bariatric surgery within 1 year prior to the screening
* Coagulation disturbances defined as (Drolz et al. 2016, Nadim et al. 2016, Stravitz et al. 2018, Green et al. 2018): fibrinogen at < 80 mg/dL and/or platelets at < 40 x 10³/mm3
* Severe hepatic encephalopathy (defined by West Haven grade > 2)
* Acute Decompensation of cirrhosis with Chronic Liver Failure Consortium Acute Decompensation (CLIF-C AD) score > 60
* Acute on Chronic liver failure (ACLF) grade 1, 2 ,3
* MELD score > 20
* Child Pugh score ≥ C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Event | up to Day 28
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Etienne SOKAL, MD, PhD, Study Chair — CSMO
Locations (13):
- Belgium (4):
  - CUB Erasme, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - University Hospital Antwerp (UZA), Edegem
  - UZ Gent, Ghent
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoana - ISUL", Sofia
  - Multiprofile hospital for active treatment (MHAT) Sofia Military Medical Academy, Sofia
  - Trakia Park Hospital, Stara Zagora
- France (2):
  - CHU Bordeaux, Bordeaux
  - Paul Brousse Hospital, Villejuif
- Spain (4):
  - Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No